CLINICAL TRIAL: NCT05529368
Title: Effect of Conventional Exercise and Tai Chi Exercise in College Students With Internet Addiction: A Randomized Clinical Trial
Brief Title: Effect of Conventional Exercise and Tai Chi Exercise on College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xueqing Zhang (Other)
Responsible Party: Sponsor-Investigator, Xueqing Zhang, Principal Investigator, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XZhang
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Internet Addiction; Exercise; Tai Chi; Randomized Clinical Trial
MeSH Terms: conditions — Internet Addiction Disorder; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional exercise group (Experimental): Participants in the conventional exercise group attended an 8-week conventional exercise program, which consisted of the track, field, ball games et al. If the participant chooses to run, the mileage shall be more than 4km and the pace shall be within 10min. The conventional exercise treatment was performed 3 times a week, 1 hour each time.
  Interventions: Behavioral: Conventional Exercise and Tai Chi Exercise interventions
- tai chi exercise group (Experimental): Participants in the tai chi exercise group attended an 8-week Yang-style 24-form tai chi training program and tai chi (8 trigrams 5 steps) which was the tai chi style most commonly adopted and studied in the literature. The tai chi exercise treatment was performed 3 times a week, 1 hour each time.
  Interventions: Behavioral: Conventional Exercise and Tai Chi Exercise interventions
- control group (No Intervention): Participants in the control group received no intervention and keep their eating and living habits.

INTERVENTIONS:
Behavioral: Conventional Exercise and Tai Chi Exercise interventions — Subjects diagnosed with IAD were randomly assigned to the exercise group, the tai chi group, or the control group. The exercise group and tai chi group received conventional exercise and tai chi for 8 weeks.
  Arms: conventional exercise group; tai chi exercise group

SUMMARY:
Internet addiction disorder (IAD) is an impulse-control disorder of Internet behavior in the absence of addictive substances. Exercise has been found to have significant advantages in improving the severity and depressive symptoms of IAD. The purpose of this study was to observe the efficacy of conventional exercise and tai chi in the treatment of Internet addiction and to observe the changes in each group. Subjects diagnosed with IAD were randomly assigned to the exercise group, the tai chi group, or the control group. The exercise group and tai chi group received conventional exercise and tai chi for 8 weeks. The Internet Addiction Test (IAT), the Pittsburgh sleep quality index (PSQI), the Zung Self-rating Depression Scale (SDS), the Zung Self-rating Anxiety Scale (SAS), and Fatigue Scale-14 (FS-14) were evaluated for all subjects at baseline and postintervention.

DETAILED DESCRIPTION:
Over the past decade, with the rapid growth and popularity of the Internet, Internet addiction (IA) has increased. Nowadays, Internet addiction disorder (IAD) has become a significant social problem, especially among teenagers and young adults. IAD is an impulse-control disorder of Internet behavior in the absence of addictive substances, its typical symptoms are involved, including tolerance, withdrawal symptoms, large amounts of time spent online, interruption of social relations, and disorder of the biological clock.

Western scholars have developed interventions for Internet addiction based on cognitive behavioral therapy (CBT). Besides applying CBT treatment, Chinese psychologists also have developed trials to apply psychoanalytic group intervention, family therapy, sports exercise prescriptions, and Naikan therapy. Physical exercise (PE) interventions are known to facilitate cerebral blood and oxygen supply, enhance brain metabolism and neurotransmitter function and improve the balance of the nervous system, which in turn helps improve physical and mental adaptability. Active physical exercise is helpful to improve the symptoms of Internet addiction. Tai chi is a mind-body exercise that originated in China. It is a form of physical and mental training combining Chinese martial arts and meditative movements involving a series of slowly performed, continuous, and rhythmic movements that put a minimal impact on the joints of the body. This study aimed to validate the use of tai chi as an alternative approach to Internet addiction and compare the effectiveness of tai chi with conventional exercise. With both primary and secondary outcome measures, the effects of tai chi and exercise on Internet addiction can be more comprehensively analyzed, which will provide a basis for its future establishment as a non-pharmacological method for the treatment of Internet addiction.

ELIGIBILITY:
Inclusion Criteria:

1. participants were diagnosed with IAD according to the Internet Addiction Test;
2. the physical activity level of participants was low;
3. participants had no history of medication or psychotherapy.

Exclusion Criteria:

1. participants had a history of severe mental illness;
2. participants had a history of drug addiction;
3. participants regularly practiced moderate-intensity exercise.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Internet Addiction Test (IAT) | 2 months
  The IAT is composed of 20 items with a 5-point scale (1 = "very rarely", 5 = "very frequently"). IAT scores range from 20 to 100, with higher scores indicating higher levels of IA. Scores over 50 indicated a tendency of IA.

SECONDARY OUTCOMES:
Pittsburgh sleep quality index (PSQI) | 2 months
  The PSQI version used in the current study was a 19-item self-report retrospective questionnaire of the past 7 days designed to measure 7 domains called component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction. Component scores range from 0 (no difficulty) to 3 (severe difficulty). PSQI scores range from 0 to 21. Scores over 7 indicated a tendency for a sleep disorder.
Zung Self-rating Depression Scale (SDS) | 2 months
  The SDS is composed of 20 items with a 4-point scale (1 = "none or a little of the time", 4 = "most or all of the time"). A standardized scoring algorithm is used to define symptoms of depression, with a total score range of 20-80. The final index score was converted by multiplying the raw score by 1.25 and then rounding off decimal places. The severity of depression was categorized according to the index score: nil depression (index score < 50), mild depression (index score 50-59), moderate depression (index score 60-69), and severe depression (index score≥70).
Zung Self-rating Anxiety Scale (SAS) | 2 months
  The SAS is composed of 20 items with a 4-point scale (1 = "none or a little of the time", 4 = "most or all of the time"). A standardized scoring algorithm is used to define symptoms of anxiety, with a total score range of 20-80. The final index score was converted by multiplying the raw score by 1.25 and then rounding off decimal places. The severity of anxiety was categorized according to the index score: nil anxiety (index score < 50), mild anxiety (index score 50-59), moderate anxiety (index score 60-69), and severe anxiety (index score≥70).
Fatigue Scale-14 (FS-14) | 2 months
  The FS-14 consists of 14 items, each of which is a fatigue-related question. The maximum total score is 14, and the higher the score, the more severe the fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Zhang, professor, Principal Investigator — Department of Epidemiology and Biostatistics, School of Public Health, Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li YY, Sun Y, Meng SQ, Bao YP, Cheng JL, Chang XW, Ran MS, Sun YK, Kosten T, Strang J, Lu L, Shi J. Internet Addiction Increases in the General Population During COVID-19: Evidence From China. Am J Addict. 2021 Jul;30(4):389-397. doi: 10.1111/ajad.13156. Epub 2021 Mar 19. PMID 33738888
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Chan AWK, Chair SY, Lee DTF, Leung DYP, Sit JWH, Cheng HY, Taylor-Piliae RE. Tai Chi exercise is more effective than brisk walking in reducing cardiovascular disease risk factors among adults with hypertension: A randomised controlled trial. Int J Nurs Stud. 2018 Dec;88:44-52. doi: 10.1016/j.ijnurstu.2018.08.009. Epub 2018 Aug 24. PMID 30195124
- [Background] Easwaran K, Gopalasingam Y, Green DD, Lach V, Melnyk JA, Wan C, Bartlett DJ. Effectiveness of Tai Chi for health promotion for adults with health conditions: a scoping review of Meta-analyses. Disabil Rehabil. 2021 Oct;43(21):2978-2989. doi: 10.1080/09638288.2020.1725916. Epub 2020 Feb 18. PMID 32070137
- [Background] He M, Yang S, Miao Y, Zhang W, Zhu D, Xu D. Four-week Tai Chi intervention decreases attention bias to drug cues in individuals with methamphetamine use disorder. Am J Drug Alcohol Abuse. 2021 Sep 3;47(5):638-648. doi: 10.1080/00952990.2021.1950745. Epub 2021 Jul 30. PMID 34325579
- [Background] Aaronson LS, Teel CS, Cassmeyer V, Neuberger GB, Pallikkathayil L, Pierce J, Press AN, Williams PD, Wingate A. Defining and measuring fatigue. Image J Nurs Sch. 1999;31(1):45-50. doi: 10.1111/j.1547-5069.1999.tb00420.x. PMID 10081212
- [Background] Li S, Wu Q, Tang C, Chen Z, Liu L. Exercise-Based Interventions for Internet Addiction: Neurobiological and Neuropsychological Evidence. Front Psychol. 2020 Jun 25;11:1296. doi: 10.3389/fpsyg.2020.01296. eCollection 2020. PMID 32670157
- [Background] Young KS. Cognitive behavior therapy with Internet addicts: treatment outcomes and implications. Cyberpsychol Behav. 2007 Oct;10(5):671-9. doi: 10.1089/cpb.2007.9971. PMID 17927535
- [Background] ZUNG WW. A SELF-RATING DEPRESSION SCALE. Arch Gen Psychiatry. 1965 Jan;12:63-70. doi: 10.1001/archpsyc.1965.01720310065008. No abstract available. PMID 14221692
- [Background] Zung WW. A rating instrument for anxiety disorders. Psychosomatics. 1971 Nov-Dec;12(6):371-9. doi: 10.1016/S0033-3182(71)71479-0. No abstract available. PMID 5172928
- [Derived] Zhang X, Yang H, Zhang K, Zhang J, Lu X, Guo H, Yuan G, Zhu Z, Du J, Shi H, Jin G, Hao J, Sun Y, Su P, Zhang Z. Effects of exercise or tai chi on Internet addiction in college students and the potential role of gut microbiota: A randomized controlled trial. J Affect Disord. 2023 Apr 14;327:404-415. doi: 10.1016/j.jad.2023.02.002. Epub 2023 Feb 6. PMID 36754096